CLINICAL TRIAL: NCT04575376
Title: Clinical Audit on Evaluation of Patient With Syncope at Asssiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MENazeer, Doctor, Assiut University
Other Study IDs: Syncope
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of commitment of resident physician to the guidelines as regard management of cases of syncope at Assiut University Children Hospital and correction of the defect that will be discovered.

DETAILED DESCRIPTION:
Definition Syncope is a transient loss of consciousness associated with inability to maintain postural tone followed by rapid and spontaneous recovery. (1)

Epidemiology About 30-50% of children have syncope at least once in their lives till adolescent period, most of them are girls, 9% is the rate of syncope in 15-17 years old adolescent group, and this rate increase to the end of adolescent period. (2)

Causes (3)

I_Neurally mediated syncope

1. Neurocardiogenic (vasovagal)

   * Emotional stress induced (pain, fear, blood phobia, etc.)
   * Orthostatic stress induced
2. Situational syncope

   * Respiratory (cough, sneeze, laugh, head turning)
   * Gastrointestinal stimulation (swallowing, defecation, postprandial)
   * Post micturition
   * Post exercise
   * Others
3. Carotid sinus syncope
4. Glossopharyngeal and trigeminal neuralgia syncope II_Cardiogenic syncope

   * Arrhythmias as Bradycardia: - sinus node dysfunction (including bradycardia/tachycardia syndrome) - atrioventricular conduction system disease Tachycardia: - supraventricular - ventricular
   * Structural heart defects as acute myocardial infarction/ischaemia, hypertrophic cardiomyopathy, cardiac masses (atrial myxoma, tumours, etc.), pericardial disease /tamponade.
   * Functional heart defects as prosthetic valve dysfunction, pulmonary hypertension.
   * Vascular heart abnormalities as aortic stenosis, congenital anomalies of coronary arteries, pulmonary embolus, acute aortic dissection.

III_ Orthostatic hypotensive syncope

* Primary autonomic disorder
* Secondary autonomic disorder
* Drug-induced orthostatic hypotension
* Hypovolemia related IV_Postural orthostatic tachycardia syndrome V_Metabolic reasons of syncope
* Hypoglycemia
* Hypoxia
* Electrolyte imbalance VI_Psychogenic syncope
* Anxiety
* Panic attack
* Depression
* Somatization VII_Drug-induced syncope
* Antihypertensives, diuretics, barbiturates, tricyclic antidepressants, alcohol, antiarrhythmics, macrolides, antihistamines, antipsychotics, MAO inhibitors, levodopa, prazosin, benzodiazepines VIII_Airway obstruction induced syncope IX_Hyperventilation-induced syncope X_Neurologic Syncope
* Cerebrovascular diseases
* Increased intracranial pressure
* Migraine

Symptoms

* The prodrome is the most important aspect of the history.
* A warm or clammy sensation, nausea, light headedness or visual changes (e.g seeing spots, grey out, tunneling)are strongly suggestive of vasovagal syndrome, other symptoms include irritability, confusion, auditory changes or dyspnea.
* The absence of prodrome raise the suspicion of a possible cardiac cause. 85%of children with vasovagal syncope has a prodrome, wheras only 40% of those with cardiac condition had a prodromal symptoms.

Palpitation and chest pain have been related to pediatric cardiac cause of syncope.(4) vasovagal syncope might also produce complex movement which raise a suspicion of epilepsy.(5)

* Most syncope is vasovagal, which is benign and doesn't require extensive investigation. The position statement presents recommendation to encourage an efficient and cost effective deposition for the many patients with a benign cause of syncope and hightlight atypical or concerning clinical findings associated with other causes of transient loss of consciousness.
* The prodrome and cirumstances around which the event occurred are the most important aspect of the history.
* Syncope occurring midexertion suggest cardiac etiology. A family history includes sudden death in the young or from unknown causes or causes that might be suspected to be other than natural can be a red flag.
* ECG is the most frequently ordered test, but the yield is low, It's recommended when patient's history isn't suggestive of vasovagal syncope and other features suggestive of cardiac cause like absence of prodrome, midexertion and family history of early life sudden death or heart diseases, abnormal physical examination or a new medication with potential cardiac cardiotoxicity.(6)

ELIGIBILITY:
Inclusion Criteria:

* all cases of syncope.

Exclusion Criteria:

-

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients with syncope who will be admitted to Assiut University Children Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Clinical audit on evaluation of a child with syncope at Assiut University children Hospital | Baseline
  Evaluation of commitment of resident physician to the guidelines as regard management of cases of syncope at Assiut University Children Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Mohie El-deen, Professor, Study Director — Asssiut University; faisal al_khateeb ahmed, Professor, Study Director — Asssiut University

REFERENCES:
- [Background] Sheldon RS, Grubb BP 2nd, Olshansky B, Shen WK, Calkins H, Brignole M, Raj SR, Krahn AD, Morillo CA, Stewart JM, Sutton R, Sandroni P, Friday KJ, Hachul DT, Cohen MI, Lau DH, Mayuga KA, Moak JP, Sandhu RK, Kanjwal K. 2015 heart rhythm society expert consensus statement on the diagnosis and treatment of postural tachycardia syndrome, inappropriate sinus tachycardia, and vasovagal syncope. Heart Rhythm. 2015 Jun;12(6):e41-63. doi: 10.1016/j.hrthm.2015.03.029. Epub 2015 May 14. No abstract available. PMID 25980576
- [Background] Johnsrude CL. Current approach to pediatric syncope. Pediatr Cardiol. 2000 Nov-Dec;21(6):522-31. doi: 10.1007/s002460010130. PMID 11050276
- [Background] Bayram AK, Pamukcu O, Per H. Current approaches to the clinical assessment of syncope in pediatric population. Childs Nerv Syst. 2016 Mar;32(3):427-36. doi: 10.1007/s00381-015-2988-8. Epub 2016 Jan 5. PMID 26732063
- [Background] Hurst D, Hirsh DA, Oster ME, Ehrlich A, Campbell R, Mahle WT, Mallory M, Phelps H. Syncope in the Pediatric Emergency Department - Can We Predict Cardiac Disease Based on History Alone? J Emerg Med. 2015 Jul;49(1):1-7. doi: 10.1016/j.jemermed.2014.12.068. Epub 2015 Mar 20. PMID 25802162
- [Background] Yilmaz S, Gokben S, Levent E, Serdaroglu G, Ozyurek R. Syncope or seizure? The diagnostic value of synchronous tilt testing and video-EEG monitoring in children with transient loss of consciousness. Epilepsy Behav. 2012 May;24(1):93-6. doi: 10.1016/j.yebeh.2012.02.006. Epub 2012 Mar 28. PMID 22459868